CLINICAL TRIAL: NCT03582709
Title: Prospective Cohort Study on Cognition and Cardiovascular Disease of Sedentary Behaviors in Children
Status: Enrolling by invitation | Type: Observational
Sponsor: CHEN Yajun (Other)
Responsible Party: Sponsor-Investigator, CHEN Yajun, Associate Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 8167120522
Record Dates: First submitted 2018-05-31; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Sedentary Behavior;Cognition;Cardiovascular-related Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood( serum,blood plasma,haemocytes)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prospective cohort study is set up to address research questions dealing with sedentary lifestyle-related events mainly including cognition and cardiovascular-related disease in children .Participants aged 7-12 years old from five primary schools in Guangzhou,Guangdong province will be recruited and followed up to evaluate the risk factors of cognition and cardiovascular-related disease. Objective measurements combined with questionnaire-data-based information on a wide range of lifestyle factors and cognition were applied in this study.

DETAILED DESCRIPTION:
There are three stages in this project.At first stage,information about socio-demographic, psychological status, physical activity,sleep and diet were collected by a multi-components questionnaire survey.The Strengths and Difficulties Questionnaire(SDQ) and Behavior Rating Inventory of Executive Function(BRIEF) were conducted at the same time. Anthropometric measurement including height, weight, waist and hip circumferences, blood pressure and fat mass were conducted.Besides,blood samples were collected to measure total cholesterol, triglycerides, high-density lipoprotein (HDL-C) and low-density lipoprotein (LDL-C).

At second stage,participants were classified for 4 subgroups as follows: Low active-high sedentary;low active-low sedentary; high active-high sedentary;high active-low sedentary by different sedentary status and physical activity levels according to the international standard. Later cardiorespiratory fitness was assessed by the 20-m shuttle run test. Accelerometer GT3X+ Actigraph with physical activity log,Combined Raven's test, a series of psychometric paradigms were measured for further studies.

At third stage,we will explore the related neuropsychological mechanism using the technology of event-related potentials (ERPs).

About 1000 participants (7-12 years old) will be prospectively followed up. The associations between sedentary lifestyle and risks for cognition and cardiovascular-related disease will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 7-12 years old
* Children with normal intelligence measured by Raven Good vision.
* Right hand.

Exclusion Criteria:

* Children with mental health and behavioral problems in this study were found to have developmental behavior disorders, such as ADHD, ASD.
* There are serious liver and kidney diseases, cardiovascular diseases, hematologic diseases or malignant tumors.

Ages: 7 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: Primary school students aged 7 to 12 in Guangzhou
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-reported physical activity and sedentary lifestyle. | 2017.01-2026.12
  Using International Physical Activity Questionnaire-Short-Chinese（IPAQ-S-C）to assess the frequency and duration of activity and sedentary lifestyle（SL） in the last 7 days .Subjects with moderate activity and vigorous activity(MVPA)≥60min/day were classified into high PA subgroup while those with MVPA<150min/week were classified into low PA subgroup according to the international standard.Subjects with SL≥gender-, age-specific 75% percentile were assigned to the high SL subgroup and< gender-, age-specific 25% percentile were assigned to the low SL subgroup.

SECONDARY OUTCOMES:
Anthropometric | 2017.01-2026.12
  Height was measured to the nearest millimeter and weight was measured to the nearest 0.1kg.Waist circumference(WC) was measured to the nearest millimeter at the level of 1cm above umbilicus with a steel tape. Body mass index(BMI) was calculated as body weight in kilograms divided by height in meters squared (kg/m2).Human body fat mass was measured by means of the bio-impedance assay ( BIA ) .Blood pressure was recorded as systolic blood pressure (SBP) and diastolic blood pressure (DBP) . Blood pressure was measured for 2 times with one-minute interval.
Biochemical indicator | 2017.01-2026.12
  Fasting blood glucose,total cholesterol, triglycerides, high-density lipoprotein (HDL-C) and low-density lipoprotein (LDL-C).
Cardiorespiratory Fitness(CRF) | 2017.01-2026.12
  CRF was assessed by the 20-m shuttle run test.Estimations of submaximal oxygen consumption (VO2max) were obtained using Leger's formulae.
Self-reported cognition | 2017.01-2026.12
  The Behavior Rating Inventory of Executive Function-Parents(BRIEF-P) examines parents' report for the frequency of "problematic" behaviors that their child displayed at home during the previous 6 months. It contains 86 items (every item chooses from three dimensions "No", "Sometimes" and "Often" ) within eight theoretically and empirically derived clinical scales that measure different aspects of executive functioning: Inhibit, Shift, Emotional Control, Initiate, Working Memory, Plan/Organize, Organization of Materials and Monitor, and three overarching composites (i.e. Behavioral Index [BRI, obtained Inhibit, Shift, Emotional Control], Metacognition Index [MI, obtained Initiate, Working Memory, Plan/Organize, Organization of Materials and Monitor] and Global Executive Composite [GEC]).The higher the score, the worse the executive function.
Objective measurement of physical activity and sedentary lifestyle. | 2017.01-2026.12
  Physical activity was measured using accelerometer GT3X+ Actigraph for 7 days continuously. The main measurement result was duration of physical activity. A wear time of ≥480 minutes/day was used as the criterion for a valid day, and ≥4 days (at least 3 weekdays and 1 weekend) were used as the criteria for a valid 7-day period of accumulated data.The cut-points for classify physical activity intensity levels are different, thus this will be specifically described in subsequent articles.
Corsi block-tapping task | 2017.01-2026.12
  Three accuracy measures were registered: The number of blocks of the longest correct sequence, the total number of correctly reproduced sequences, and the product of these two measures.
Stroop task | 2017.01-2026.12
  Response accuracy and reaction time(RT) were collected to assess behavioral performance.
Wisconsin Card Sorting Test(WCST) | 2017.01-2026.12
  Children with poor executive function exhibited a higher error rate and slower reaction times.
Combined Raven's Test | 2017.01-2026.12
  The correct number of questions is calculated to reflect intelligence level.(Level 1: a test standard score of high intelligence equal to or greater than 95% of the constant module of the same age.Level 2: good intelligence is between 75% and 95%.Level 3:average intelligence is between 25% and 75%. Level 4:the low level of intelligence is between 5% and 25%.Level 5: mental retardation is less than 5%)
Event-related potentials | 2018.09-2026.12
  Assessing cognition using the Event-Related Potentials (ERPs) methodology of certain early and late ERPs (i.e. P1, N1, N2, P2, P3).EEG activity was collected during the cognitive tasks from 64 electrode sites to derive and assess separately the ERPs amplitude and latency measures.

REFERENCES:
- [Derived] Lv Y, Cai L, Zeng X, Gui Z, Lai L, Tan W, Chen Y. Association between weekend catch-up sleep and executive functions in Chinese school-aged children. J Clin Sleep Med. 2020 Aug 15;16(8):1285-1293. doi: 10.5664/jcsm.8494. PMID 32279704
- [Derived] Lv Y, Cai L, Gui Z, Zeng X, Tan M, Wan N, Lai L, Lu S, Tan W, Chen Y. Effects of physical activity and sedentary behaviour on cardiometabolic risk factors and cognitive function in children: protocol for a cohort study. BMJ Open. 2019 Oct 31;9(10):e030322. doi: 10.1136/bmjopen-2019-030322. PMID 31676650